CLINICAL TRIAL: NCT00640094
Title: Randomized, Double-blind, Parallel-group, Placebo-controlled Study of Melatonin as an Adjunct in Patients With Acute myocaRdial Infarction Undergoing Primary Angioplasty
Brief Title: The Melatonin Adjunct in the Acute myocaRdial Infarction Treated With Angioplasty
Acronym: MARIA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Alberto Domínguez Rodríguez (Other)
Responsible Party: Sponsor-Investigator, Alberto Domínguez Rodríguez, MD, PhD, FESC, Fundación Canaria Rafael Clavijo para la Investigación Biomédica
Organization: Fundación Canaria Rafael Clavijo para la Investigación Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005-000821-49
Record Dates: First submitted 2008-03-12; First posted 2008-03-20 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Acute Myocardial Infarction
Keywords: Melatonin; Acute myocardial infarction; Primary angioplasty
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Melatonin (Experimental): Melatonin: intravenous infusion and intracoronary bolus
  Interventions: Drug: melatonin
- B: Placebo of melatonin (Placebo Comparator): Placebo: intravenosus infusion and intracoronary bolus
  Interventions: Drug: melatonin

INTERVENTIONS:
Drug: melatonin — Patients will receive a total intravenous melatonin dose of 12 mg + intracoronary melatonin dose of 2 mg. The intravenous dose will be distributed in a volume of 50 ml of a isotonic and sterile solution and administered by intravenous infusion during 60 minutes. The intracoronary dose will be distributed in a volume of 10 ml of a isotonic and sterile solution and administered as a bolus.
  Other Names: 5-methoxy-tryptamine

SUMMARY:
Background: Experimental studies have documented the beneficial effects of the endogenously produced antioxidant, melatonin, in reducing tissue damage and limiting cardiac pathophysiology in models of experimental ischemia-reperfusion. Melatonin confers cardioprotection against ischemia-reperfusion injury most likely through its direct free radical scavenging activities and its indirect actions in stimulating antioxidant enzymes. These actions of melatonin permit it to reduce molecular damage and limit infarct size in experimental models of transient ischemia and subsequent reperfusion.

Study design: The Melatonin Adjunct in the acute myocaRdial Infarction treated with Angioplasty (MARIA) trial is a prospective, randomized, double-blind, placebo-controlled, phase 2 study of the intravenous administration of melatonin. The primary efficacy end point of this study is to determine whether melatonin treatment reduces infarct size determined by cardiac magnetic resonance 5-7 days post-reperfusion. Other secondary end points will be the clinical events occurring within the first year: death, sustained ventricular arrhythmias, resuscitation from cardiac arrest, cardiogenic shock, heart failure, major bleedings , stroke, need for revascularization, recurrent ischemia, re-infarctions and rehospitalization; and changes in left ventricular ejection fraction from baseline to 4 months of follow-up.

Implications: The MARIA trial tests a novel pharmacologic agent, melatonin, in patients with acute myocardial infarction and the hypothesis that it will confer cardioprotection against ischemia-reperfusion injury. If successful, the finding would support the use of melatonin in therapy of ischemic-reperfusion injury of the heart.

DETAILED DESCRIPTION:
See article for more detailed description: Contemporary Clinical Trials 28 (2007) 532-539

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years.
2. Having experienced continuous ischemic (cardiac) symptoms for at least 20 minutes.
3. Having onset of symptoms of qualifying acute myocardial infarction within the past 6 hours and be expected to undergo primary angioplasty.
4. Having an electrocardiogram indicative of an acute ST segment -elevation myocardial infarction showing:

   > 2 mm ST segment elevation in 2 anterior or lateral leads; or > 2 mm ST segment elevation in 2 inferior leads coupled with ST depression in 2 contiguous anterior leads for a total ST deviation of > 8 mm; or new left bundle branch block with at least 1 mm concordant ST elevation.
5. Being willing to provide informed consent (informed consent may be provided by a legally authorized representative if the patient is not able to provide it according to local ethical standards).
6. Being willing and able to be followed for at least 3 months for evaluation.

Exclusion Criteria:

A patient will be ineligible for study entry if he/she meets any of the following criteria:

1. prehospital thrombolysis,
2. Killip class IV on admission,
3. known history of prior myocardial infarction,
4. known history of renal failure,
5. history of severe allergic reaction,
6. history of autoimmune diseases,
7. pregnancy,
8. severe concurrent illness with reduced short-term prognosis,
9. inability to give informed consent and
10. participation in another study within the past 30 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2013-05; Primary Completion 2016-03 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Infarct size | 5-7 days post-reperfusion
  The primary efficacy end point in this study is to determine whether melatonin treatment reduces infarct size (percentage of total myocardial necrotic mass) by cardiac magnetic resonance

SECONDARY OUTCOMES:
Major cardiac events: Death, sustained ventricular arrhythmias, resuscitation from cardiac arrest, cardiogenic shock, heart failure, major bleedings, stroke, need for revascularization, recurrent ischemia, re-infarctions and re-hospitalization. | within the first year
Changes in left ventricular ejection fraction evaluated by cardiac magnetic resonance | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Dominguez-Rodriguez, MD, PhD, FESC, Principal Investigator
Locations (3):
- Spain (3):
  - Hospital General Universitario Santa Lucia, Cartagena, Murcia
  - University Hospital of Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Universitario Marqués de Valdecilla, Santander

REFERENCES:
- [Result] Dominguez-Rodriguez A, Abreu-Gonzalez P, Garcia-Gonzalez MJ, Kaski JC, Reiter RJ, Jimenez-Sosa A. A unicenter, randomized, double-blind, parallel-group, placebo-controlled study of Melatonin as an Adjunct in patients with acute myocaRdial Infarction undergoing primary Angioplasty The Melatonin Adjunct in the acute myocaRdial Infarction treated with Angioplasty (MARIA) trial: study design and rationale. Contemp Clin Trials. 2007 Jul;28(4):532-9. doi: 10.1016/j.cct.2006.10.007. Epub 2006 Oct 17. PMID 17123867